CLINICAL TRIAL: NCT02455973
Title: Interdisciplinary Intervention Effectiveness on Motivational Approach in Lifestyle Modification in Adolescents With Overweight and Obesity
Brief Title: Interdisciplinary Intervention With Motivational Approach in Adolescents With Overweight and Obesity.
Acronym: MERC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MERC
Record Dates: First submitted 2015-04-25; First posted 2015-05-28 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Overweight
Keywords: obesity; overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Heart Disease Risk Factors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transtheoretical model of change (Experimental): In this type of intervention, the focus will be the development of skills through educational activities on health based on interdisciplinary motivational strategies.
  Interventions: Behavioral: Lifestyle modification and cardiovascular risk
- Health information (Placebo Comparator): In this type of intervention, the focus will be the development of skills through educational activities on health using the pedagogy of transmission.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Lifestyle modification and cardiovascular risk — Group meetings will be performed in the presence of a member of the nursing staff, physiotherapy, nutrition and psychology. The meetings are weekly, lasting 1 hour and 45 minutes. In the first 1 hour and 15 minutes will be addressed health issues related to lifestyle modification (self-care, healthy eating and physical activity) using the fundamentals of motivational interviewing technique. All topics will be focused on the major cardiovascular risk factors considered modifiable.Likewise, it is envisaged to include a time of physical activity (30 minutes) oriented in conjunction with the research team. Run in: There will be a meeting with the parents in order to inform them about the participation of children in the program and guide them about the procedures of the research protocol.
  Arms: Transtheoretical model of change
Behavioral: Health Education — The meetings will be weekly with 45 minutes duration on a schedule of lectures about cardiovascular risk
  Arms: Health information

SUMMARY:
This study is a randomized clinical trial with two interventions: control group and intervention interdisciplinary group, without cross-over.

Control Group (CG): In this type of intervention, the focus will be the development of skills through educational activities on health using the pedagogy of transmission.

Interdisciplinary Intervention Group (IG): In this type of intervention, the focus will be the development of skills through educational activities on health that provide the development of autonomy and empowerment for behavior change, based on interdisciplinary motivational strategies. All topics will be focused on the major cardiovascular risk factors considered modifiable.

The staff is trained to the techniques of motivational interviewing and transtheoretical model of change and the health issues related to the modification of lifestyle.

So this interdisciplinary intervention with adolescents seeks to measure the result of an educational proposal using the techniques of motivational interviewing and transtheoretical model of change, for all professionals involved independent training in health issues related approach to lifestyle modification and the inclusion of family in this process.

DETAILED DESCRIPTION:
This study is a randomized clinical trial with two interventions: control group and intervention interdisciplinary group, without cross-over.

Interventions will take place at the Rehabilitation Hospital São Lucas Center (CR), will have 12 sessions for each of the following ways:

Control Group (CG): In this type of intervention, the focus will be the development of skills through educational activities on health using the pedagogy of transmission. The meetings will be weekly with 45 minutes duration on a schedule of lectures about cardiovascular risk factors and prevention.The sample is 60 adolescents with overweight or obesity.

Interdisciplinary Intervention Group (IG): In this type of intervention, the focus will be the development of skills through educational activities on health that provide the development of autonomy and empowerment for behavior change, based on interdisciplinary motivational strategies. Therefore, group meetings will be performed in the presence of a member of the nursing staff, physiotherapy, nutrition and psychology. The meetings are weekly, lasting 1 hour and 45 minutes. In the first 1 hour and 15 minutes will be addressed health issues related to lifestyle modification (self-care, healthy eating and physical activity) using the fundamentals of motivational interviewing technique. All topics will be focused on the major cardiovascular risk factors considered modifiable.

The staff is trained to the techniques of motivational interviewing and transtheoretical model of change and the health issues related to the modification of lifestyle. During the sessions the team members address the health issue so that the knowledge of a professional complements the other. At the same time occur the integration of knowledge between these professionals from different areas aiming to encourage teens to lifestyle modification based on the techniques of motivational interviewing and transtheoretical model of change. Likewise, it is envisaged to include a time of physical activity (30 minutes) oriented in conjunction with the research team. This activity aims to motivate adolescents to include other physical activity sessions during the week.

So this interdisciplinary intervention with adolescents seeks to measure the result of an educational proposal using the techniques of motivational interviewing and transtheoretical model of change, for all professionals involved independent training in health issues related approach to lifestyle modification and the inclusion of family in this process.

Run in: There will be a meeting with the parents of the IG and CG (separately) in order to inform them about the participation of children in the program and guide them about the procedures of the research protocol.

ELIGIBILITY:
Inclusion Criteria:

Adolescents between 15 and 18 years with BMI ≥ 85th percentile.

Exclusion Criteria:

Provide absolute contraindication for physical activity for musculoskeletal, neurological, vascular problems (intermittent claudication), lung and heart; presence of diagnosis of severe psychiatric disorders and / or presence of significant cognitive impairments;pregnant women; diagnosis of Diabetes mellitus type I.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) measured by height and weight and taking the z score. | Measured after three months at the end of intervention
  Reduction of at least 0.5 percentile point in body mass index (BMI) measured by height and weight and taking the z score.

SECONDARY OUTCOMES:
Abdominal circumference measured by waist circumference in cm | Measured after three months at the end of intervention
  Reduction of at least 5% abdominal circumference measured by waist circumference in cm
Dietary aspects as measured by healthy eating index (IAS) | Measured after three months at the end of intervention
  Improves 5% of the Diet quality measured by healthy eating index (IAS)
Capacity cardiopulmonary measured by VO2 max | Measured after three months at the end of intervention
  Increase 5% in capacity cardiopulmonary measured by VO2 max
Blood pressure measured by the blood pressure measurement | Measured after three months at the end of intervention
  Reduced at least 7% in systolic blood pressure measured by the blood pressure measurement
Plasma triglycerides measured by the blood sample | Measured after three months at the end of intervention
  Reduction of at least 20% of the plasma triglycerides measured by the blood sample
Plasma HDL cholesterol measured by the blood sample | Measured after three months at the end of intervention
  Increase of at least 5% of the plasma HDL cholesterol measured by the blood sample
Total cholesterol and LDL measured by the blood sample | Measured after three months at the end of intervention
  Reduction of at least 5% in total cholesterol and LDL measured by the blood sample
Glycemic profile assessed by fasting glucose | Measured after three months at the end of intervention
  Glycemic profile is expected to be reduced by at least 5% at the end of the intervention assessed by fasting glucose
Readiness for change measured by the readiness ruler to physical exercise | Measured after three months at the end of intervention
  Increase of one point in the continuous variable readiness to change for performing physical exercise measured by the readiness ruler to physical exercise
Readiness for change measured by the readiness ruler to physical nutrition | Measured after three months at the end of intervention
  Increase of one point in the continuous variable readiness to change for performing physical nutrition measured by the readiness ruler to physical exercise

CONTACTS AND LOCATIONS:
Overall Officials: Margareth da Silva Oliveira, PHD, Principal Investigator — Pontifical Catholic University of Rio Grande do Sul
Locations (1):
- Pontifical Catholic University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Miller WR, Rose GS. Toward a theory of motivational interviewing. Am Psychol. 2009 Sep;64(6):527-37. doi: 10.1037/a0016830. PMID 19739882
- [Background] Prochaska JO, DiClemente CC, Norcross JC. In search of how people change. Applications to addictive behaviors. Am Psychol. 1992 Sep;47(9):1102-14. doi: 10.1037//0003-066x.47.9.1102. PMID 1329589
- [Background] Velasquez M; Maurer GG; Crouch C; DiClemente CC. Group treatment for substance abuse: a stages-of- change therapy manual. New York: The Guilford Press, 2001. 222 p.
- [Background] Miller WR; Rollnick S. Motivational Interviewing, Second Edition: Preparing People for Change.New York, NY: The Guilford Press, 2002. 482 p.
- [Derived] Zanatta LB, Heinzmann-Filho JP, Vendrusculo FM, Campos NE, Oliveira MDS, Feoli AMP, Gustavo ADS, Donadio MVF. Effect of an interdisciplinary intervention with motivational approach on exercise capacity in obese adolescents: a randomized controlled clinical trial. Einstein (Sao Paulo). 2020;18:eAO5268. doi: 10.31744/einstein_journal/2020ao5268. Epub 2020 May 18. PMID 32428066